CLINICAL TRIAL: NCT04498351
Title: Evaluation of Magnesium Sulfate in Combination With Dexmedetomidine As Adjuvants to Levobupivacaine for Augmenting Analgesia and Anesthesia in Ultrasound Guided Spermatic Cord Block For Testicular Sperm Extraction Surgery
Brief Title: Magnesium Sulfate in Combination With Dexmedetomidine As Adjuvants to Levobupivacaine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: N-19-2020
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Spermatic Cord Block
Keywords: Spermatic Cord Block; Magnesium Sulfate; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: Following skin sterilization and local anesthetic infiltration of the superficial tissues, an echogenic 22-G block needle is inserted in-plane to the ultrasound beam in a cranial-to-caudal direction the spermatic cord in short axis and directed towards the deferent duct, contralateral to the testicular artery. The needle tip was advanced to become contact with the deferent. Correct location of the needle tip was confirmed by injecting 0.5-1 ml to see the local anesthetic spreading around the deferent duct. A total of 18ml levobupivacaine 0.5% are then injected into the spermatic cord block .
  The procedure is repeated on the contralateral side.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Prospective randomized double blinded clinical study on humans
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cotrol group (Placebo Comparator)
  Interventions: Drug: Control Test
- dexmedetomidine group (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- magnesium sulphate group (Active Comparator)
  Interventions: Drug: magnesium sulphate
- dexmedetomidine and magnesium sulphate group (Active Comparator)
  Interventions: Drug: Dexmedetomidine and magnesium sulphate

INTERVENTIONS:
Drug: Control Test — Spermatic cord block by18ml levobupivacaine 0.5% plus 2 ml normal saline in total volume of 20 ml.
  The procedure is repeated on the contralateral side.
  Arms: cotrol group
Drug: Dexmedetomidine — Spermatic cord block by total of 18ml levobupivacaine 0.5% plus 1 μg/kg dexmedetomidine in 2 ml in total volume of 20 ml The procedure is repeated on the contralateral side.
  Arms: dexmedetomidine group
Drug: Dexmedetomidine and magnesium sulphate — Spermatic cord block by total of 18ml levobupivacaine 0.5% plus 1 μg/kg dexmedetomidine and 100 mg magnesium sulphate in 2 ml in total volume of 20 ml .
  The procedure is repeated on the contralateral side.
  Arms: dexmedetomidine and magnesium sulphate group
Drug: magnesium sulphate — Spermatic cord block by total of 18ml levobupivacaine 0.5% plus 100 mg magnesium sulphate in 2 ml in total volume of 20 ml
  Arms: magnesium sulphate group

SUMMARY:
Using the spermatic cord block has been of great advantage, as it has been cost saving, efficient technique whether used inon its own or combination with a sedative or . Furthermore, it provides minimal cardiac risks, early case ambulation, satisfactory postoperative pain control, as well as a reduced hospital stay and cost. one of the major drawbacks of spermatic cord block is being a single injection technique, leading to a short postoperative analgesia duration. So, to overcome this flaw some adjuvants were proven to prolong the analgesia duration as Dexmetedomidine (Dex), and magnesium.

DETAILED DESCRIPTION:
The technique of the spermatic cord block was first described in the 1960s by Earle AS.Using the spermatic cord block has been of great advantage, as it has been cost saving, efficient technique whether used inon its own or combination with a sedative or . Furthermore, it provides minimal cardiac risks, early case ambulation, satisfactory postoperative pain control, as well as a reduced hospital stay and cost. one of the major drawbacks of spermatic cord block is being a single injection technique, leading to a short postoperative analgesia duration. So, to overcome this flaw some adjuvants were proven to prolong the analgesia duration as Dexmetedomidine (Dex), and magnesium.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 60 years.
* ASA I-II.
* Undergoing Testicular Sperm Extraction Surgery.
* BMI from 18.5 to 30 kg/m2

Exclusion Criteria:

* Patient refusal
* Contraindications to regional anesthesia (bleeding disorders e.g. INR>1.5, PC<70%, platelet count<100 × 109, use of any anti-coagulants, local infection, etc.).
* Known allergy to local anesthetics.
* ASA III-IV.
* Patients aged less than 18 or more than 60.
* Body mass index >35.
* Patients with difficulty in evaluating their level of pain.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — the operation only in male
Enrollment: 130 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Time from injection of LA to the first postoperative analgesic request | UP TO 1 HOURE
  (duration of the block).

SECONDARY OUTCOMES:
heart rate | up to 24 hours
  beat/min
VAS | up to 24 hours
  0 No Pain 1-3 Mild Pain (nagging, annoying, interfering little with ADLs) 4-6 Moderate Pain (interferes significantly with ADLs) 7-10 Severe Pain (disabling; unable to perform ADLs)
perform SCAB | UP TO 1 HOURE
  The mean time needed to perform SCAB
total nalbuphine consumption | up to 24 hours
  total nalbuphine consumption
Incidence of complications | up to 24 hours
  complications
mean arterial blood pressure | up to 24 hours
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: mohamad abdulfatah, MD, Principal Investigator — lecture
Locations (1):
- Faculty of Medicine, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
still working